CLINICAL TRIAL: NCT01389544
Title: Investigation of the Effect of Multiple Doses of Danoprevir/Ritonavir on Methadone in Subjects on Stable Methadone Maintenance Therapy (MMT)
Brief Title: A Study on the Interaction Between Danoprevir/Ritonavir and Methadone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NP25644
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Methadone; Ritonavir

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: danoprevir; Drug: methadone; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — 200 mg daily (100 mg q12h) orally, Days 1-10
Drug: methadone — stable maintenance therapy: 20-120 mg daily single oral morning dose
Drug: ritonavir — 200 mg daily (100 mg q12h) orally, Days 1-10

SUMMARY:
This multicenter, open-label study will assess the effect of multiple doses of danoprevir/ritonavir on steady-state pharmacokinetics of methadone. Subjects on stable methadone maintenance therapy (20 - 120 mg daily as single oral morning dose) will receive danoprevir 100 mg orally twice daily and ritonavir 100 mg orally twice daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 - 65 years of age, inclusive
* Subjects must be on a stable methadone maintenance regimen (20 to 120 mg/day) for the treatment of opiate addiction for at least 30 days prior to screening and should be on a stable dose for at least 14 days prior to Day -1
* Body weight >/= 50 kg
* Body mass index (BMI) 18.0 - 32.0 kg/m2
* Females of childbearing potential and males with female partners of childbearing potential must agree to use 2 forms of non-hormonal contraception during the study and for 90 days after the last study drug administration

Exclusion Criteria:

* Pregnant or lactating women and male partners of women who are pregnant or lactating
* Symptoms of methadone withdrawal at screening, on Day -2 or Day -1
* Inadequate venous access
* History or evidence of any clinically significant disease or disorder, except for drug abuse or dependence
* Positive test for alcohol or drugs of abuse at screening and up to Day -2 (with the exception of methadone)
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol); alcohol consumption will be prohibited during study confinement and for at least 48 hours before screening, dosing and each scheduled visit
* Positive for hepatitis B, hepatitis C or HIV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effect of danoprevir/ritonavir on steady state pharmacokinetics (area under the concentration - time curve (AUC)) of methadone | 10 days

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Anaheim, California
  - Overland Park, Kansas